CLINICAL TRIAL: NCT07018960
Title: "Multicenter Registry for Chest Wall Reconstruction Surgery Using Custom Dynamic Prostheses PRODIPET"
Brief Title: "Multicenter Registry for Chest Wall Reconstruction Using Custom Dynamic Prostheses (PRODIPET)"
Acronym: PRODIPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Hospital Universitario de la Ribera (Unknown); Hospital de Cruces (Other); Hospital Universitario Insular de Gran Canaria. Las Palmas de GG. Spain (Unknown); University Hospital of Girona Dr. Josep Trueta (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRODIPET
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Chest Wall Tumors; Post-traumatic Syndrome; Malignant Bone Tumor of Chest Wall
Keywords: Chest wall tumors; Chest wall reconstruction; Custom 3D-Printed Titanium Prostheses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Dynamic Chest Wall Reconstruction with Patient-Specific 3D-Printed Titanium Prostheses" (Experimental)
  Interventions: Procedure: Chest wall reconstruction with 3D printed titan custom prothesis

INTERVENTIONS:
Procedure: Chest wall reconstruction with 3D printed titan custom prothesis — Dynamic Chest Wall Reconstruction with Patient-Specific 3D-Printed Titanium Prostheses"
  1. Intervention Overview
  A custom-designed, 3D-printed titanium prosthesis is surgically implanted to reconstruct chest wall defects following oncologic resection or traumatic injury. The prosthesis is engineered to:
  Restore structural integrity of the thoracic cavity Preserve physiological chest wall dynamics during respiration Provide long-term biomechanical stability

SUMMARY:
PRODIPET Study Summary

Title: Multicenter Registry for Chest Wall Reconstruction Using Custom 3D-Printed Titanium Prostheses

Purpose

The PRODIPET study evaluates the safety and effectiveness of personalized, dynamic titanium prostheses for reconstructing the chest wall after:

Tumor resection (e.g., sarcomas, lung cancer). Severe trauma (e.g., multiple rib fractures). Traditional methods (metal plates, mesh) often lack flexibility, potentially causing pain or breathing difficulties. This study tests 3D-printed titanium implants designed to mimic natural rib movement, improving function and comfort.

Study Design

Type: Multicenter, ambispective (retrospective + prospective data).

Duration:

Prospective: 24 months (Jan 2024-Jan 2026). Follow-up: 12 months per patient (final analysis by 2027). Centers: Major Spanish hospitals (Ramón y Cajal/Madrid, La Ribera/Alzira, Cruces/Baracaldo, Insular/Las Palmas).

Key Goals

Assess short/mid-term outcomes (pain, breathing, complications). Compare results across patients/surgical techniques. Improve future prosthesis designs. Who Can Participate?

Inclusion:

Adults (18+) needing chest wall reconstruction. Signed consent for anonymized data sharing.

Exclusion:

Titanium allergies. Participation in conflicting studies. Patient Experience

Pre-Surgery:

CT scan creates a custom 3D prosthesis (made by Osteobionix® using Ti6AL4V-ELI titanium).

Surgery:

Surgeons implant the prosthesis, anchoring it to ribs/sternum.

Follow-Up:

Evaluations at discharge, 1/6/12 months (in-person or phone). Measures: Pain, lung function, imaging (X-ray/CT), complications (e.g., infection, implant failure).

Privacy & Ethics

Data is anonymized and stored securely (REDCap system). Complies with European General Data Protection Regulation (EU GDPR) and Spanish data protection laws.

Patients may withdraw anytime. For Healthcare Providers

Collaboration: Open to thoracic surgeons/researchers. Data Access: Centralized via REDCap; analyzed by the coordinating team. Publications: Multicenter results will be published first; individual centers may later share their data.

Why This Matters

Addresses a gap in evidence for dynamic prostheses, which may offer:

Better breathing mechanics vs. rigid materials. Fewer long-term complications (e.g., breakage). Could standardize best practices for complex reconstructions. Contact

Lead Coordinator: Dr. Nicolás Moreno Mata (Hospital Ramón y Cajal, Madrid). Email: nicolas.moreno.hrc@gmail.com | Phone: +34 647 609 363.

Key Takeaways:

Patients/Families: Learn if custom prostheses improve recovery. Providers: Contribute to advancing surgical options. Researchers: Access multicenter data on innovative implants.

DETAILED DESCRIPTION:
Here's a detailed yet accessible description of the PRODIPET study:

**PRODIPET Study: A Comprehensive Multicenter Investigation into 3D-Printed Titanium Chest Wall Reconstruction**

**Background and Rationale** Chest wall defects resulting from tumor resections or traumatic injuries present significant surgical challenges. Traditional reconstruction methods using rigid materials like methylmethacrylate or steel plates often compromise respiratory mechanics and patient comfort. The PRODIPET study examines an innovative solution: patient-specific, 3D-printed titanium prostheses designed to replicate natural chest wall dynamics.

**Study Design and Methodology**

This national multicenter registry combines:

* Retrospective data: Cases from participating centers where titanium prostheses were previously implanted
* Prospective data: New cases enrolled over a 24-month period (January 2024-January 2026)

**Technical Innovation**

The prostheses are:

* Custom-designed using preoperative CT scans
* Manufactured via electron beam melting of Ti6AL4V-ELI titanium powder
* Engineered to provide:

  * Anatomical precision
  * Dynamic flexibility mimicking natural rib movement
  * Reduced imaging artifacts for better postoperative monitoring

**Clinical Protocol**

1. Preoperative Phase:

   * Multidisciplinary evaluation (surgeons, radiologists, engineers)
   * Virtual surgical planning using 3D reconstruction
   * Prosthesis fabrication by Osteobionix® (2-3 week turnaround)
2. Surgical Phase:

   * Resection of affected chest wall segment
   * Implantation of custom prosthesis
   * Fixation to remaining ribs/sternum
3. Postoperative Follow-up:

   * Standardized evaluations at:

     * Hospital discharge
     * 1 month
     * 6 months
     * 12 months
   * Assessments include:

     * Pulmonary function tests
     * Pain scales (VAS)
     * CT imaging
     * Quality of life questionnaires

**Data Collection and Management**

* Secure REDCap database hosted by EJIE (Informatic Society of Basque Government, IT)
* Comprehensive variables tracked:

  * Demographic data
  * Surgical details (operative time, blood loss)
  * Prosthesis characteristics (size, fixation method)
  * Complication rates
  * Functional outcomes

**Participant Protection**

* CEIm (ethical committee)-approved protocol (Hospital Ramón y Cajal Ethics Committee)
* GDPR-compliant data handling
* Two-tier identification system:

  1. Local centers maintain identifiable information
  2. Central registry uses anonymized codes
* Right to withdraw without penalty

**Scientific Objectives**

Primary:

* Determine prosthesis durability (12-month failure rate)
* Assess restoration of pulmonary function

Secondary:

* Identify optimal candidates for this technique
* Establish complication profiles
* Compare outcomes across surgical centers
* Refine prosthesis design parameters

**Clinical Significance**

This study addresses critical gaps in thoracic reconstruction by:

* Providing real-world evidence for a novel technology
* Establishing standardized protocols
* Creating a benchmark for future innovations
* Potentially improving quality of life for patients requiring extensive chest wall resection

**Collaborative Structure**

* Coordinating Committee: 4 lead thoracic surgeons
* Participating Centers: Open to all Spanish hospitals meeting criteria
* Industry Partner: Osteobionix® (device fabrication only, no data access)

**Dissemination Plan**

* Interim analysis at 12 months
* Final results publication anticipated 2027
* Data sharing policy:

  * Coordinating committee controls primary dataset
  * Participating centers may publish local data after multicenter publication

This rigorous, patient-focused investigation represents a significant advancement in thoracic surgical care, combining cutting-edge engineering with clinical expertise to improve outcomes for patients with complex chest wall defects.

ELIGIBILITY:
Inclusion Criteria

Patients must meet ALL of the following:

• Age: ≥18 years

Clinical Indication:

* Requires chest wall reconstruction due to:
* Oncologic resection (primary tumors, metastases)
* Traumatic injury (flail chest, severe rib fractures)
* Post-infection/post-radiation defects
* Defect Characteristics:
* Involves ≥2 ribs or sternum with instability
* Minimum defect size: 5 cm in largest dimension
* Surgical Plan:
* Scheduled for reconstruction with 3D-printed custom titanium prosthesis
* Consent: Willing to provide informed consent for:
* Surgery
* Data collection
* Follow-up evaluations
* Exclusion Criteria

Patients will be excluded if ANY of the following apply:

* Medical Contraindications:
* Active systemic infection (e.g., sepsis)
* Severe cardiopulmonary disease (FEV₁ <30% predicted)
* Uncorrectable coagulopathy (INR >1.5)
* Technical Limitations:
* Inadequate soft tissue coverage for prosthesis
* Vertebral column involvement requiring complex fixation
* Material Incompatibility:
* Known hypersensitivity to titanium alloys
* Study Logistics:
* Participation in another conflicting clinical trial
* Inability to complete follow-up (e.g., no fixed address)
* Ethical Considerations:
* Pregnancy (due to elective CT scan requirements)
* Prisoners or cognitively impaired patients without legal guardians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Respiratory Outcomes: Change from Baseline in Spirometric Parameters Following 3D-Printed Titanium Chest Wall Reconstruction | From enrollment to the end of treatment at 1 year
  *Measured via spirometry according to ATS/ERS /The American Thoracic Society/European respiratory society) standards at 30 days and 1 year postoperatively*
Change from Preoperative Baseline in Forced Vital Capacity (FVC) | From enrollment to the end of treatment at 1 year
  *Measured via spirometry according to ATS/ERS standards at 30 days and 1 year postoperatively*
Change from Preoperative Baseline in FEV₁/FVC Ratio | From enrollment to the end of treatment at 1 year
  Calculated from spirometry results at 30 days and 1 year postoperatively
Change from Preoperative Baseline in Peak Expiratory Flow (PEF) | From enrollment to the end of treatment at 1 year
  Measured via spirometry at 30 days and 1 year postoperatively
Change from Preoperative Baseline in Forced Expiratory Flow 25-75% (FEF₂₅-₇₅%) | From enrollment to the end of treatment at 1 year
  Measured via spirometry at 30 days and 1 year postoperatively

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital de Cruces, Cruces, Basque Country
  - Complejo Hospitalario Universitario Insular, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Josep Trueta, Barcelona, Catalonia
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario de La Ribera, Alzira, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://osteobionix.com